CLINICAL TRIAL: NCT00445458
Title: A Phase 1/2 Study of HKI-272 in Combination With Paclitaxel in Subjects With Solid Tumors and Breast Cancer
Brief Title: A Phase 1/2 Study of HKI-272 (Neratinib) in Combination With Paclitaxel (Taxol) in Subjects With Solid Tumors and Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3144A1-203 / B1891014
Record Dates: First submitted 2007-03-08; First posted 2007-03-09 (Estimated); Results first posted 2018-05-09 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Advanced Breast Cancer; Advanced Malignant Solid Tumors; Breast Neoplasms
Keywords: cancer; HKI-272; neratinib; paclitaxel; Taxol; breast cancer; Nerlynx
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — neratinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- HKI-272 dose level 1 (Experimental): Part 1: Subjects with solid tumors receiving HKI-272 (neratinib) 160 mg daily by mouth in combination with paclitaxel 80 mg/m^2 weekly IV.
  Interventions: Drug: HKI-272; Drug: Paclitaxel
- HKI-272 dose level 2 (Experimental): Part 1: Subjects with solid tumors receiving HKI-272 (neratinib) 240 mg daily by mouth in combination with paclitaxel 80 mg/m^2 weekly IV.
  Interventions: Drug: HKI-272; Drug: Paclitaxel
- HKI-272 expanded MTD cohort, arm A (Experimental): Part 2: Subjects with metastatic breast cancer who have not received more than 1 prior cytotoxic chemotherapy treatment regimen for metastatic disease receiving HKI-272 (neratinib) 240 mg daily by mouth in combination with paclitaxel 80 mg/m^2 weekly IV.
  Interventions: Drug: HKI-272; Drug: Paclitaxel
- HKI-272 expanded MTD cohort, arm B (Experimental): Part 2: Subjects with metastatic breast cancer who have not received more than 3 prior cytotoxic chemotherapy treatment regimen for metastatic disease receiving HKI-272 (neratinib) 240 mg daily by mouth in combination with paclitaxel 80 mg/m^2 weekly IV.
  Interventions: Drug: HKI-272; Drug: Paclitaxel

INTERVENTIONS:
Drug: HKI-272
  Other Names: Neratinib
Drug: Paclitaxel

SUMMARY:
The purpose of this study is to learn whether it is safe and effective to administer HKI-272 (neratinib) in combination with paclitaxel in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for both parts of clinical trial:

* Good performance status
* Normal ejection fraction
* Adequate cardiac, kidney, and liver function
* Adequate blood counts
* At least one measurable target lesion
* Negative pregnancy test for female subjects

Inclusion Criteria for Part 1 Only:

- Pathologically confirmed solid tumor not curable with available standard therapy

Inclusion Criteria for Part 2 Only:

* Pathologically confirmed breast cancer
* HER2 positive tumor
* Prior treatment with Herceptin

Exclusion Criteria:

Exclusion criteria for both parts of clinical trial:

* Major surgery, radiotherapy, chemotherapy or investigational agents within two weeks of treatment day 1
* Subjects with bone or skin as the only site of disease
* Active central nervous system metastases
* Significant cardiac disease or dysfunction
* Significant gastrointestinal disorder
* Inability or unwillingness to swallow HKI-272 capsules
* Prior exposure to HKI-272 or other HER2 targeted agents, except trastuzumab (Part 2 only). Prior lapatinib is permitted in arm B of part 2.
* Treatment with a taxane within 3 months of treatment day 1
* Grade 2 or greater motor or sensory neuropathy
* Pregnant or breast feeding women
* Known hypersensitivity to paclitaxel or Cremophor EL
* Prior treatment with anthracyclines with cumulative dose of >400 mg/m^2
* Any other cancer within 5 years with the exception of contralateral breast cancer, adequately treated cervical carcinoma in situ, or adequately treated basal or squamous cell carcinoma of the skin

Exclusion Criteria for Part 2 Only:

- More than 1 (arm A) or 3 (arm B) prior cytotoxic chemotherapy regimen for metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-09-11 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2018-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (32):
- United States (8):
  - Scripps, Clinic General, La Jolla, California
  - Moores UC San Diego Cancer Center, La Jolla, California
  - Sharp Memorial Hospital, San Diego, California
  - Boston University Medical Center, Boston, Massachusetts
  - Mid-Michigan Physicians-HOS Division, Lansing, Michigan
  - Oncology Care Associates, Saint Joseph, Michigan
  - Columbia University Medical Center, New York, New York
  - CTRC at The University of Texas Health Science Center, San Antonio, Texas
- Belgium (4):
  - Institut Jules Bordet Unite du Chimiotherapie, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge Campus Maria's Voorzienigheid (MV), Kortrijk
  - Oncologisch Centrum GZA - Location St Augustinus, Wilrijk
- Princess Margaret Hospital University Health Network, Toronto, Ontario, Canada
- China (6):
  - The Hospital Affiliated Academy Military Medical Science, Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Tianjin Union Medicine Center Department of Oncology, Tianjin, Tianjin Municipality
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking Union Medical College Hospital of Chinese Academy of Medical Sciences, Beijing
- Hong Kong (3):
  - UNIMED Medical Institute, Hong Kong
  - Department of Medicine, Queen Mary Hospital, Hong Kong
  - Department of Surgery Queen Mary Hospital, Hong Kong
- India (4):
  - Jehangir Clinical Development Centre, Jehangir Hospital Premises, Pune, Maharashtra
  - M.M.F. Joshi Hospital & Ratna Memorial Hospital, Pune, Maharashtra
  - Tata Memorial Hospital, Mumbai, Parel
  - Birla Cancer Centre, S.M.S. Medical College & Hospital, Jaipur, Rajasthan
- Poland (2):
  - Wojewodzki Szpital Specjalistyczny im. Ludwika Rydygiera, Oddzial Onkologii, Krakow
  - Oddzial Chemioterapii Centrum Onkologii Ziemii Lubelskiej, Lublin
- South Korea (2):
  - Yonsei University Health System - Severance Hospital, Seoul
  - Asan Medical Center, Division of Oncology, Department of Internal Medicine, Seoul
- Ukraine (2):
  - City Multifield Clinical Hospital #4 Department of chemotherapy, Dnipropetrovs'k State Medical Academy, Chair of Oncology and Medical Radiology, Dnipropetrovsk
  - State Oncological Regional Treatment and Diagnostic Center Department of chemotherapy, Lviv

REFERENCES:
- [Derived] Chow LW, Xu B, Gupta S, Freyman A, Zhao Y, Abbas R, Vo Van ML, Bondarenko I. Combination neratinib (HKI-272) and paclitaxel therapy in patients with HER2-positive metastatic breast cancer. Br J Cancer. 2013 May 28;108(10):1985-93. doi: 10.1038/bjc.2013.178. Epub 2013 Apr 30. PMID 23632474

RESULTS

PARTICIPANT FLOW:
Groups:
- Neratinib 160 mg + Paclitaxel 80 mg/m2: Neratinib 160 mg qd + Paclitaxel 80 mg/m2 IV on days 1, 8, and 15 of a 28 day cycle.
- Neratinib 240 mg + Paclitaxel 80 mg/m2: Neratinib 240 mg qd + Paclitaxel 80 mg/m2 IV on days 1, 8, and 15 of a 28 day cycle.
- Arm A Neratinib (MTD) + Paclitaxel 80 mg/m2: Neratinib (MTD) qd + Paclitaxel 80 mg/m2 on days 1, 8, and 15 of a 28 day cycle for subjects with not more than 1 prior cytotoxic chemotherapy treatment regimen for metastatic disease.
- Arm B Neratinib (MTD) + Paclitaxel 80 mg/m2: Neratinib (MTD) + Paclitaxel 80 mg/m2 on days 1, 8, and 15 of a 28 day cycle for subjects with not more than 3 prior cytotoxic chemotherapy treatment regimen for metastatic disease.
Period: Overall Study
Arm/Group | Neratinib 160 mg + Paclitaxel 80 mg/m2 | Neratinib 240 mg + Paclitaxel 80 mg/m2 | Arm A Neratinib (MTD) + Paclitaxel 80 mg/m2 | Arm B Neratinib (MTD) + Paclitaxel 80 mg/m2
Started | 3 | 5 | 71 | 31
Completed | 0 | 0 | 3 | 3
Not Completed | 3 | 5 | 68 | 28
Not completed — Disease Progression | 3 | 4 | 54 | 27
Not completed — Withdrawal by Subject | 0 | 0 | 7 | 0
Not completed — Adverse Event | 0 | 0 | 3 | 0
Not completed — Death | 0 | 1 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1
Not completed — Surgery | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Arm A Neratinib (MTD) + Paclitaxel: Neratinib (MTD) + Paclitaxel 80 mg/m2 on days 1, 8, and 15 of a 28 day cycle for subjects with not more than 1 prior cytotoxic chemotherapy treatment regimen for metastatic disease
- Arm B Neratinib (MTD) + Paclitaxel: Neratinib (MTD) + Paclitaxel 80 mg/m2 on days 1, 8, and 15 of a 28 day cycle for subjects with not more than 3 prior cytotoxic chemotherapy treatment regimen for metastatic disease
- Total: Total of all reporting groups
Arm/Group | Neratinib 160 mg + Paclitaxel 80 mg/m2 | Neratinib 240 mg + Paclitaxel 80 mg/m2 | Arm A Neratinib (MTD) + Paclitaxel | Arm B Neratinib (MTD) + Paclitaxel | Total
Number analyzed (Participants) | 3 | 5 | 71 | 31 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (14.57) | 49.6 (11.72) | 49.2 (10.10) | 51.4 (8.50) | 50.0 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 71 | 31 | 105
  Male | 2 | 3 | 0 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 48 | 25 | 77
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 0 | 3 | 22 | 5 | 30
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity Incidence of Neratinib in Combination With Paclitaxel
Description: Dose Limiting Toxicity in subjects with solid tumors treated with neratinib, administered daily, in combination with paclitaxel 80 mg/m² IV on days 1, 8, and 15 of a 28 day cycle.
Time Frame: From first dose date through day 28
Population: Safety population of Study Part 1. Treated set including patients eligible for MTD determination.
Measure: Count of Participants; unit: Participants
Groups:
- Neratinib 160 mg + Paclitaxel 80 mg/m²: Neratinib 160 mg qd + Paclitaxel 80 mg/m² IV on days 1, 8, and 15 of a 28 day cycle.
- Neratinib 240 mg + Paclitaxel 80 mg/m²: Neratinib 240 mg qd + Paclitaxel 80 mg/m² IV on days 1, 8, and 15 of a 28 day cycle.
Arm/Group | Neratinib 160 mg + Paclitaxel 80 mg/m² | Neratinib 240 mg + Paclitaxel 80 mg/m²
Number analyzed (Participants) | 3 | 5
Participants | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose
Description: Maximum Tolerated Dose (MTD) of neratinib, daily, in combination with paclitaxel 80 mg/m², intravenous at days 1, 8, and 15, associated with the dose limiting toxicity data.
Time Frame: From first dose date through day 28.
Population: Safety population of Study Part 1. Treated set including patients eligible for MTD determination.
Measure: Number; unit: mg
Groups:
- Part 1. Neratinib + Paclitaxel 80 mg/m²: Daily Administration of Neratinib in combination with Paclitaxel 80 mg/m2 IV on days 1, 8, and 15 of a 28 day cycle.
Arm/Group | Part 1. Neratinib + Paclitaxel 80 mg/m²
Number analyzed (Participants) | 8
mg | 240

3. Primary Outcome: Objective Response Rate
Description: Subjects with partial response (PR) or complete response (CR) with ERBB2 positive breast cancer treated at the maximum tolerated dose (MTD) of neratinib in combination with paclitaxel, per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v.1.0: CR, disappearance of all target lesions; PR, >=30% decrease in the sum of the longest diameter of target lesions; and no progressive disease (PD) for non-target lesions, and no new lesions.
Time Frame: From first dose date to progression or last tumor assessment, up to 140 weeks
Population: All subjects, in Study part 2 evaluable population, who met the inclusion/exclusion criteria, received at least 2 weeks of neratinib and at least 2 doses of paclitaxel, and underwent at least 1 post-Baseline tumor assessment. Subjects who died or had symptomatic deterioration before the first scheduled post-Baseline tumor assessment were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm A Neratinib (MTD) + Paclitaxel: Neratinib (MTD) + Paclitaxel 80 mg/m² on days 1, 8, and 15 of a 28 day cycle for subjects with not more than 1 prior cytotoxic chemotherapy treatment regimen for metastatic disease.
- Arm B Neratinib (MTD) + Paclitaxel: Neratinib (MTD) + Paclitaxel 80 mg/m² on days 1, 8, and 15 of a 28 day cycle for subjects with not more than 3 prior cytotoxic chemotherapy treatment regimens for metastatic disease.
Arm/Group | Arm A Neratinib (MTD) + Paclitaxel | Arm B Neratinib (MTD) + Paclitaxel
Number analyzed (Participants) | 68 | 31
percentage of participants | 70.6 [58.3 to 81.0] | 77.4 [58.9 to 90.4]

4. Secondary Outcome: Maximum Plasma Concentration of Neratinib
Description: Maximum plasma concentration of neratinib; after each dosing of neratinib on Cycle 1 of Day 15, blood samples taken at regular time points.
Time Frame: Samples taken at 0 hour and at 1, 2, 4, 6, 8, and 24 hours postdose on Day 15 of Cycle 1, and 1 predose sample on Day 1 in Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Neratinib 160 mg + Paclitaxel 80 mg/m²: Neratinib 160 mg, once a day, orally, in combination with paclitaxel 80 mg/m², IV, given on days 1, 8, and 15 of a 28 day cycle.
- Neratinib 240 mg + Paclitaxel 80 mg/m²: Neratinib 240 mg, once a day, orally, in combination with paclitaxel 80 mg/m², IV, given on days 1, 8, and 15 of a 28 day cycle.
Arm/Group | Neratinib 160 mg + Paclitaxel 80 mg/m² | Neratinib 240 mg + Paclitaxel 80 mg/m²
Number analyzed (Participants) | 3 | 94
ng/mL | 66.78 (25) | 80.42 (55)

5. Secondary Outcome: Area Under the Concentration-time Curve 0-24
Description: Area under the concentration-time curve of neratinib; after each dosing of neratinib on Cycle 1 of Day 15, blood samples taken at regular time points.
Time Frame: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Neratinib 160 mg + Paclitaxel 80 mg/m² | Neratinib 240 mg + Paclitaxel 80 mg/m²
Number analyzed (Participants) | 3 | 94
h*ng/mL | 684 (92) | 1274 (61)

ADVERSE EVENTS:
Time Frame: From first dose through 28 days after last dose, up to 140 weeks.
Groups:
- Neratinib 160 mg + Paclitaxel 80 mg/m2: Neratinib 160 mg qd + Paclitaxel 80 mg/m2 on days 1, 8, and 15 of a 28 day cycle.
- Neratinib 240 mg+ Paclitaxel 80 mg/m2: Neratinib 240 mg qd + Paclitaxel 80 mg/m2 on days 1, 8, and 15 of a 28 day cycle.
- Arm A Neratinib 240 mg (MTD) + Paclitaxel 80 mg/m2: Neratinib (MTD) qd + Paclitaxel 80 mg/m2 on days 1, 8, and 15 of a 28 day cycle for subjects with not more than 1 prior cytotoxic chemotherapy treatment regimen for metastatic disease
- Arm B Neratinib 240 mg (MTD) + Paclitaxel 80 mg/m2: Neratinib (MTD) qd + Paclitaxel 80 mg/m2 on days 1, 8, and 15 of a 28 day cycle for subjects with not more than 3 prior cytotoxic chemotherapy treatment regimen for metastatic disease
Arm/Group | Neratinib 160 mg + Paclitaxel 80 mg/m2 | Neratinib 240 mg+ Paclitaxel 80 mg/m2 | Arm A Neratinib 240 mg (MTD) + Paclitaxel 80 mg/m2 | Arm B Neratinib 240 mg (MTD) + Paclitaxel 80 mg/m2
Serious Adverse Events (participants affected / at risk) | 1/3 | 4/5 | 27/71 | 4/31
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 70/71 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib 160 mg + Paclitaxel 80 mg/m2 (N=3) | Neratinib 240 mg+ Paclitaxel 80 mg/m2 (N=5) | Arm A Neratinib 240 mg (MTD) + Paclitaxel 80 mg/m2 (N=71) | Arm B Neratinib 240 mg (MTD) + Paclitaxel 80 mg/m2 (N=31)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 6 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Fungaemia (Infections and infestations) | 0 | 0 | 1 | 0
Malaria (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib 160 mg + Paclitaxel 80 mg/m2 (N=3) | Neratinib 240 mg+ Paclitaxel 80 mg/m2 (N=5) | Arm A Neratinib 240 mg (MTD) + Paclitaxel 80 mg/m2 (N=71) | Arm B Neratinib 240 mg (MTD) + Paclitaxel 80 mg/m2 (N=31)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 24 | 11
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 29 | 15
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 37 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 4 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 3 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 5 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 8 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 10 | 3
Constipation (Gastrointestinal disorders) | 1 | 0 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 65 | 29
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 8 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 5 | 3
Gingival ulceration (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 5 | 0
Nausea (Gastrointestinal disorders) | 0 | 4 | 26 | 7
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 13 | 5
Vomiting (Gastrointestinal disorders) | 0 | 3 | 20 | 4
Asthenia (General disorders) | 0 | 0 | 13 | 7
Axillary pain (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 16 | 6
Generalised oedema (General disorders) | 0 | 0 | 0 | 2
Local swelling (General disorders) | 0 | 0 | 1 | 2
Malaise (General disorders) | 1 | 2 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 6 | 2
Oedema peripheral (General disorders) | 0 | 2 | 13 | 5
Pain (General disorders) | 1 | 0 | 2 | 1
Pyrexia (General disorders) | 0 | 0 | 18 | 4
Drug hypersensitivity (Immune system disorders) | 1 | 2 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 4 | 1
Influenza (Infections and infestations) | 0 | 1 | 6 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 7 | 2
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 9 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 10 | 5
Alanine aminotransferase increased (Investigations) | 0 | 0 | 10 | 6
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 9 | 4
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 10 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 16 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 6 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 7 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 8 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 7 | 4
Headache (Nervous system disorders) | 0 | 0 | 10 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1 | 36 | 17
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 2
Dysuria (Renal and urinary disorders) | 1 | 0 | 3 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 16 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 9 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 5 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 37 | 12
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 7 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 21 | 8
Hot flush (Vascular disorders) | 0 | 1 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less